CLINICAL TRIAL: NCT00458497
Title: Effect of Holofiber Socks and Bedding on Pain and Quality of Sleep in Subjects With Chronic Foot Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Hologenix, LLC (Industry)
Responsible Party: Ian Gordon, M.D., Ph.D, VA Long Beach Health Care System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #788
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Diabetic Neuropathy; Arthritis; Peripheral Arterial Disease; Plantar Fasciitis
Keywords: Holofiber; chronic foot pain; sleep quality
MeSH Terms: conditions — Diabetic Neuropathies; Arthritis; Peripheral Arterial Disease; Fasciitis, Plantar; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects will be given 3 pairs of socks (subjects with foot pain only) and bedding (mattress pad)fabricated from 1.8 dernier polyethylene terephthalate (PET) fabric to which Holofiber particles have been added during fiber manufacture.
  Interventions: Device: Holofiber fabric
- 2 (Placebo Comparator): Subjects will be given 3 pairs of socks (subjects with foot pain only) and bedding (mattress pad)fabricated from 1.8 dernier polyethylene terephthalate (PET) fabric.
  Interventions: Device: PET fabric

INTERVENTIONS:
Device: Holofiber fabric — Subjects will be given 3 pairs of socks (subjects with foot pain only) and bedding (mattress pad)fabricated from 1.8 dernier polyethylene terephthalate (PET) fabric to which Holofiber particles have been added during fiber manufacture.
  Arms: 1
Device: PET fabric — Subjects will be given 3 pairs of socks (subjects with foot pain only) and bedding (mattress pad)fabricated from 1.8 dernier polyethylene terephthalate (PET)fabric.
  Arms: 2

SUMMARY:
This study is designed to assess the effects of socks and bedding materials on foot pain, the level of blood oxygen existing in the feet and quality of sleep in subjects who have chronic foot pain from either diabetic neuropathy or other conditions, e.g., peripheral arterial disease, regenerative joint disease). The three main hypotheses to be tested are: 1)compared to placebo socks, subjects wearing Holofiber socks experience reduction in foot pain, 2)compared to placebo bedding, subjects sleeping in beds lined with a Holofiber mattress pad experience improved quality of sleep and 3) compared to placebo socks, subjects who wear Holofiber socks will have increased blood oxygenation levels in their feet.

DETAILED DESCRIPTION:
Holofiber is a patented process for adding micron sized optically active quartz, aluminum oxide and titanium oxide particles to polymer yarns. It is believed that the Holofiber particles increase skin illumination such that pigments and other enzymes are activated, leading to increased blood flow and oxygenation of the skin and neighboring soft tissues. Previous clinical trials have demonstrated approximately a 7% increase in skin oxygen levels with the use of Holofiber gloves and socks, compared to gloves and socks fabricated from identical polymer fiber lacking the optical particles. Numerous anecdotal reports from patients with chronic foot and arm pain indicate wearing Holofiber garments for even a few days leads to dramatic improvement in many different painful conditions. Similarly, many subjects with chronic sleep disturbances have reported improved quality of sleep using Holofiber bedding. The current study is designed to 1) substantiate the ability of Holofiber socks to alleviate chronic pain resulting from diabetic neuropathy and other chronic foot disorders, 2) determine if Holofiber bedding improves quality of sleep and 3) determine if Holofiber socks increase blood oxygenation levels in the feet after wear.

Subjects who give informed consent and meet the study inclusion and exclusion criterial will undergo a brief medical history and physical examination, including monofilament testing for sensory neuropathy and measurement of blood pressure in all four extremities using Doppler ultrasound, and will answer a panel of questionnaires that assess pain and sleep quality. Spouses or partners of eligible subjects will similarly be consented to fill out the questionnaires related to sleep if they share the same bed with the participating subject. Subjects and spouses/partners will be asked to return one week later to complete the same questionnaires, at which time subjects will be randomized (double-blind) to receive either Holofiber or placebo socks and bedding materials. Subjects will be instructed to use the socks and bedding material exclusively for two weeks. Subjects and spouses/partners will return at three and four weeks for follow-up with repeat questionnaires at each visit. At Visit 4, subjects will have their feet photographed using a Hyperspectral camera to identify blood oxygenation before and after wearing the Holofiber and placebo socks. Once the final set of photographs has been taken, the visit is ended and the patients participation is concluded.

ELIGIBILITY:
Inclusion Criteria SUBJECTS WITH DIABETIC NEUROPATHY:

* Presence of diabetic neuropathic pain with score of 3 or higher on the McGill Short Form Pain Survey
* Presence of sensory neuropathy with monofilament (Semmes-Weinstein) testing, as defined as failure to sense the filament in 2 locations (out of six total) on a least one foot.
* Previous diagnosis of diabetes (type II) as well as diabetic neuropathy by a physician
* Age greater or equal to 21

Exclusion Criteria SUBJECTS WITH DIABETIC NEUROPATHY:

* Presence of significant peripheral arterial disease in either lower extremity (abi greater than 0.9 bilaterally)
* Skin ulceration on either foot or limb threat from infection or vascular disease at study enrollment
* Inability to comply with study procedures or give informed consent
* Women of child bearing potential
* Spouse/partner is a women of child bearing potential and you share the same bed
* Non-ambulatory status
* Inability to comply with study restrictions on changing sleeping or pain medication
* Severe psychiatric or medical disorder that would affect compliance
* Known allergy to PET or Dacron

Inclusion Criteria SUBJECTS WITHOUT DIABETIC NEUROPATHY:

* Chronic foot or angle pain with a score of 3 or higher on the McGill Short Form Pain Scale
* Absence of sensory neuropathy with monofilament (Semmes-Weinstein) testing, as defined as ability to sense the filament in 6 locations (out of 6 total) on both feet
* The presence of a condition that causes chronic foot pain such as arthritis, peripheral arterial disease, plantar fasciitis, or other conditions not related to diabetic neuropathy, previously diagnosed by a health care provider
* Age greater to or equal to 21

Exclusion Criteria SUBJECTS WITHOUT DIABETIC NEUROPATHY:

* Presence of significant peripheral arterial disease in either lower extremity (abi less than or equal to 0.5 in either extremity)
* Skin ulceration on either foot or limb threat from infection or vascular disease at study enrollment
* Inability to comply with study procedures or give informed consent
* Women of child bearing potential
* Spouse/partner is a women of child bearing potential and you share the same bed
* Non-ambulatory status
* Inability to comply with study restrictions on changing sleeping or pain medication
* Severe psychiatric or medical disorder that would affect compliance
* Previous diagnosis of neuropathy affecting lower extremities
* Known allergy to PET or Dacron

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Significant differences between the average scores from the two pre-randomization questionnaire sets and the two post-randomization questionnaire sets. | four weeks
Oxygenation levels of blood in the feet will be compared between Holofiber and placebo socks at several time points using standard nonparametric t-test statistics. | Baseline photos of feet without socks; immediately afer baseline photos, Holofiber sock placed on one foot, placebo sock placed on the other foot; second photos with socks one hour later; final photos with socks four hours later

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gordon, M.D., Ph.D., Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Derived] York RM, Gordon IL. Effect of optically modified polyethylene terephthalate fiber socks on chronic foot pain. BMC Complement Altern Med. 2009 Apr 22;9:10. doi: 10.1186/1472-6882-9-10. PMID 19386127
- See also: Southern California Institute for Research and Education website — http://www.scire-lb.org